CLINICAL TRIAL: NCT02188238
Title: Effect of Active Ingredients in Oral Health Products on the in Vitro Structure of the Acquired Salivary Pellicle.
Brief Title: Effect of Oral Health Ingredients on the Acquired Salivary Pellicle
Status: Completed | Type: Observational
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: IFR01/2014
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: saliva; protein; oral health; film; pellicle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Saliva Sample Collection: Collection of stimulated whole mouth saliva . Whole mouth saliva is collected through stimulation by inert gum, and collecting saliva in a sterile tube.
  Interventions: Other: Saliva Sample Collection

INTERVENTIONS:
Other: Saliva Sample Collection — Saliva samples will be collected from healthy volunteers recruited locally. Stimulated whole mouth saliva is collected through stimulation by inert gum, and collecting the saliva by gently spitting into a sterile tube.
  Other Names: Stimulated Whole Mouth Saliva

SUMMARY:
The aim of this study is to help us understand how saliva forms a thin film inside the surfaces of the mouth which is known as the salivary pellicle, and how this film helps to protect our teeth from decay. We know that the thickness and physical properties (viscosity and mechanical strength) of the salivary pellicle influences:-

* How we chew and sense the structure of food in our mouth.
* How we digest the food and extract nutrients from it.
* Protection against tooth decay and infection.

However, studies have only recently established the different proteins within the pellicle. The effects of oral care products (e.g. toothpaste, mouthwash etc.) and ingredients they contain on pellicle formation and removal remain poorly understood. Therefore we need to understand how the formation of the salivary pellicle is controlled by ingredients it comes into contact with such as those from food and oral hygiene products (e.g. toothpaste and mouthwash).

In this study, we are asking volunteers to provide samples of saliva. We will take the saliva samples back to our labs and measure how they form films under different conditions and determine the influence of ingredients from oral hygiene on the film forming properties. We will also measure the protein content of the saliva sample to see how this affects pellicle formation. Eventually, this information together with knowledge from other studies, should lead to the development of more effective oral hygiene products.

DETAILED DESCRIPTION:
Saliva contains many proteins and components that contribute to film formation, and we know that saliva forms complex, structured films on surfaces. The mucosal salivary layer, comprises of a mobile layer of saliva and an immobile film of salivary proteins adsorbed onto oral epithelial cells, the "mucosal pellicle". The salivary film is thin (10-100 µm), extremely viscoelastic and aids lubrication, influences the sensory perception of food in the mouth and maintains oral health. The apparent viscoelastic and coating properties of saliva are in fact mainly due to the formation of an incredibly strong, viscoelastic film at surfaces and interfaces. The solution viscosity of saliva is actually close to that of water at high shear rates, but the interfacial viscosity is more than 10,000 times greater than water, which completely dominates the physical properties of the salivary film as a whole. This complex structure is driven by molecular scale interactions and is thought to be responsible for the film forming properties of saliva. What is still unclear are the fundamental physical and molecular mechanisms underlying the film forming properties of saliva. Although the viscous and lubricating properties of saliva have often been assigned to mucins, it appears that isolated mucins do not impart the same lubrication properties as they do in whole saliva. Other proteins such as statherin have been implicated in enhancing boundary lubrication. The molecular composition of salivary proteins and the presence of ions appear to be all important in forming the salivary film. For example, parotid saliva which contains no mucin is still highly lubricating probably due to its highly visco-elastic surface layer.

The mucosal pellicle can be mimicked in vitro by adsorbing salivary proteins onto model surfaces to form interfacial films and has been shown to be highly lubricating. The presence of polyphenols has been shown to reduce the lubricity of these surface films and correlate well with their sensory properties. At the Quadram Institute Bioscience (QIB) we have over 20 years' experience studying proteins at interfaces and surfaces, in particular how competitive adsorption at interfaces of proteins with surfactants and other surface-active components can affect the composition, structure and stability of the interface, and how this controls the functionality of the system as a whole. This was applied in a collaborative study on interfacial salivary films with Kings College London, where we demonstrated the highly visco-elastic nature of the salivary film and the critical importance of calcium ions in its formation.

Leading up to this project, the recent postgraduate (PhD) student project at QIB demonstrated that added calcium can strengthen the salivary pellicle, and that the formation of the pellicle was a two stage process involving small, surface active proteins in the primary stage, and larger mucin proteins in the later stage. The study also demonstrated that reducing pH reduced the integrity of the pellicle, which helps us to understand the role of the pellicle in preventing acid erosion, and that the addition of various active ingredients from toothpaste and mouthwash would remove certain proteins from the pellicle, depending on the type of active ingredient and the surface on which the pellicle was formed. We would like to extend this project to look at how these active ingredients in mouthwash and toothpaste affect the structure of the pellicle, and if any combinations of these ingredients have any additional effect.

Therefore our hypothesis is that active ingredients from toothpastes and mouthwashes can be used to control the structure of the salivary pellicle through their interactions with either the surface that the pellicle is adsorbed to, or with the proteins in the pellicle itself.

Understanding these changes to the structure and properties of the salivary film could then help us understand how the pellicle and the active ingredients protect teeth against decay and disease.

ELIGIBILITY:
Inclusion Criteria:

* Apparently Healthy
* Age: 18 - 65y
* Gender: Male or Female
* Non-smokers
* There are no restrictions regarding dietary habits

Exclusion Criteria:

* have known diabetes
* have any medical history of Tuberculosis or Hepatitis
* have depressed or elevated blood pressure measurements (<90/50 or <95/50 if symptomatic or >160/100).
* are currently undergoing any medical investigations
* have undergone any dental or mouth surgery, or tongue piercing within the last six weeks
* take any medication which may affect saliva production
* have any ongoing or chronic dental or mouth problems that may influence saliva composition
* have jaw or chewing problems which may be exacerbated by the saliva collection procedure
* are related to someone in the study team i.e. spouse, partner or immediate family member
* are pregnant, planning to become pregnant, or are currently breastfeeding.
* are not prepared to remove any tongue "piercings" prior to the saliva collection procedure.
* If results of the clinical screening which indicate, or are judged by the Human Nutrition Unit's (HNU) Medical Advisor to be indicative of, a health problem which compromise the well-being of the volunteer if they participated, or which would affect the study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparently healthy volunteers from the local community able to donate saliva samples
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Thickness (Depth, nm) of Salivary Films Adsorbed Onto Solid Surfaces | Within 4 hours of saliva collection
  The principal output is to determine how ingredients in oral hygiene products affect the way that the protein in saliva forms films on surfaces similar to those found inside the mouth. We will determine the main physical properties of the film such as thickness (nm), adsorbed mass (ng/cm^2), density (ng/cm^3) measured by adsorbing whole mouth saliva onto solid silica surfaces and measuring the above properties of the film using Dual Polarisation Interferometry and a Quartz Crystal Microbalance. The effect of ingredients from oral hygiene products on the above measured parameters will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Wilde, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute Bioscience, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Background] Ash A, Burnett GR, Parker R, Ridout MJ, Rigby NM, Wilde PJ. Structural characterisation of parotid and whole mouth salivary pellicles adsorbed onto DPI and QCMD hydroxyapatite sensors. Colloids Surf B Biointerfaces. 2014 Apr 1;116:603-11. doi: 10.1016/j.colsurfb.2013.10.024. Epub 2013 Nov 12. PMID 24269053
- [Background] Ash A, Ridout MJ, Parker R, Mackie AR, Burnett GR, Wilde PJ. Effect of calcium ions on in vitro pellicle formation from parotid and whole saliva. Colloids Surf B Biointerfaces. 2013 Feb 1;102:546-53. doi: 10.1016/j.colsurfb.2012.08.048. Epub 2012 Sep 7. PMID 23104024
- See also: Link to IFR homepage — http://www.ifr.ac.uk
- See also: Principal Investigator homepage — http://www.ifr.ac.uk/profile/peter-wilde.asp